CLINICAL TRIAL: NCT00537927
Title: The Effect of Mesh Fixation Technique on Postoperative Pain in Laparoscopic Correction of Incisional and Ventral Abdominal Wall Hernias.
Brief Title: LACH-Trial: LAparoscopic Correction of Hernia
Acronym: LACH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ziekenhuisgroep Twente (Other)
Responsible Party: EB Wassenaar, MD, Ziekenhuisgroep Twente
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P05-28
Record Dates: First submitted 2007-10-01; First posted 2007-10-02 (Estimated); Last update posted 2009-02-18 (Estimated); Status verified 2009-01

CONDITIONS: Incisional Hernia; Ventral Hernia
Keywords: laparoscopic correction; ventral and incisional hernia; mesh fixation; postoperative pain
MeSH Terms: conditions — Incisional Hernia; Hernia, Ventral; Pain, Postoperative | interventions — Melanocyte-Stimulating Hormones; Lavsan; Polyglactin 910

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 0 (Active Comparator): fixation of mesh with a single crown of tacks and absorbable sutures
  Interventions: Procedure: laparoscopic correction of hernia with mesh
- 1 (Active Comparator): fixation of mesh with a double crown of tacks and no sutures
  Interventions: Procedure: laparoscopic correction of hernia with mesh
- 2 (Active Comparator): fixation of mesh with a single crown of tacks and non-absorbable sutures
  Interventions: Procedure: laparoscopic correction of hernia with mesh

INTERVENTIONS:
Procedure: laparoscopic correction of hernia with mesh — Correction of hernia with mesh and fixation of mesh using one of the arms.
  Other Names: DualMesh; Mersilene; Vicryl; ProTack; Suture Passer

SUMMARY:
Method of fixation of the mesh in laparoscopic incisional / ventral hernia repair might influence the degree of postoperative pain.

The study hypothesis is that there is no difference in postoperative pain between different methods to fix the mesh in laparoscopic incisional / ventral hernia repair.

DETAILED DESCRIPTION:
One of the complications in laparoscopic incisional / ventral hernia repair is postoperative pain. Method of fixation of the mesh in laparoscopic incisional / ventral hernia repair might influence the degree of this postoperative pain. Fixation of the mesh might also influence other outcome parameters such as return to preoperative activities, costs and recurrence rate.

The study hypothesis is that there is no difference in postoperative pain when comparing three commonly used mesh fixation techniques in laparoscopic incisional / ventral hernia repair.

ELIGIBILITY:
Inclusion Criteria:

* Non-acute incisional hernia of the abdominal wall or ventral hernia of the abdominal wall
* Informed consent
* Elective surgery

Exclusion Criteria:

* < 18 years and > 80 years
* Prednison > 15 mg/24hr, started more than 2 weeks prior to surgery
* Chronical cough (severe COPD etc)
* Ascites
* Peritoneal dialysis
* Current abdominal infection
* Complete loss of abdominal domain due to hernia (diameter more than 10 cm?)
* Re-laparoscopic correction of ventral hernia

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 215 (Actual)
Dates: Start 2005-08; Primary Completion 2008-10 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Assessment of postoperative pain | one year

SECONDARY OUTCOMES:
Quality of life | one year
Overall satisfaction | one year
Postoperative stay | one month
Per- and postoperative morbidity | one month
Recurrence | Three years

CONTACTS AND LOCATIONS:
Overall Officials: Eelco B Wassenaar, MD, Principal Investigator — Ziekenhuisgroep Twente; Srjdan Rakic, MD, PhD, Study Director — Ziekenhuisgroep Twente
Locations (1):
- Ziekenhuisgroep Twente, Almelo, Netherlands

REFERENCES:
- [Background] Goodney PP, Birkmeyer CM, Birkmeyer JD. Short-term outcomes of laparoscopic and open ventral hernia repair: a meta-analysis. Arch Surg. 2002 Oct;137(10):1161-5. doi: 10.1001/archsurg.137.10.1161. PMID 12361426
- [Background] DeMaria EJ, Moss JM, Sugerman HJ. Laparoscopic intraperitoneal polytetrafluoroethylene (PTFE) prosthetic patch repair of ventral hernia. Prospective comparison to open prefascial polypropylene mesh repair. Surg Endosc. 2000 Apr;14(4):326-9. doi: 10.1007/s004640020013. PMID 10790548
- [Background] LeBlanc KA. Laparoscopic incisional and ventral hernia repair: complications-how to avoid and handle. Hernia. 2004 Dec;8(4):323-31. doi: 10.1007/s10029-004-0250-5. PMID 15235939
- [Background] Heniford BT, Park A, Ramshaw BJ, Voeller G. Laparoscopic repair of ventral hernias: nine years' experience with 850 consecutive hernias. Ann Surg. 2003 Sep;238(3):391-9; discussion 399-400. doi: 10.1097/01.sla.0000086662.49499.ab. PMID 14501505
- [Derived] Wassenaar E, Schoenmaeckers E, Raymakers J, van der Palen J, Rakic S. Mesh-fixation method and pain and quality of life after laparoscopic ventral or incisional hernia repair: a randomized trial of three fixation techniques. Surg Endosc. 2010 Jun;24(6):1296-302. doi: 10.1007/s00464-009-0763-1. Epub 2009 Dec 24. PMID 20033726